CLINICAL TRIAL: NCT06511453
Title: Remote Self-Administered Acupressure for Pain Management in Patients With Sickle Cell Disease
Brief Title: Acupressure in Patients With Sickle Cell Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Ying Wang, Assistant Professor of Anesthesia, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10056b
Record Dates: First submitted 2024-07-10; First posted 2024-07-22 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Pain; Acupressure; Inner Eyelid Imaging
MeSH Terms: conditions — Anemia, Sickle Cell; Pain | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Usual Care + Acupressure (Experimental): Participants will continue ongoing usual care and administer self-acupressure treatment.
  Interventions: Device: Acupressure (using AcuWand or pencil eraser)
- Usual Care Only (No Intervention)

INTERVENTIONS:
Device: Acupressure (using AcuWand or pencil eraser) — The acupressure procedure will consist of medium-deep pressure as tolerated at each assigned point applied in a circular motion. Subjects will be trained in the appropriate performance of the treatment at all points and complete the first treatment under supervision. Acupressure treatment will last for 2-3 minutes per point and be administered remotely every other day for 5 weeks.
  Acupressure will be performed using a tool (AcuWand) and a pencil (the pencil's eraser head will be used as an alternative/backup tool) will be provided to help participants apply the right amount of pressure on the appropriate points on their bodies. In the event AcuWand/pencil is not available, participants can use fingers/thumbs for self-acupressure.
  Arms: Usual Care + Acupressure

SUMMARY:
The proposed research is to determine the clinical efficacy and neurobiological mechanisms of acupressure analgesia in patients with sickle cell disease (SCD).

DETAILED DESCRIPTION:
This study will help the investigators learn whether acupressure, a non-pharmacological alternative treatment approach, can help manage pain in patients with sickle cell disease. Acupressure involves the application of pressure stimulation at specific acupoints on the body. Acupressure may help relieve pain and is used for a wide variety of pain conditions. Participation in this study will consist of remote self-administered treatment every other day over 5 weeks, followed by 6 months of remote follow-up visits. During participation, subjects will: 1) receive detailed instruction on locating treatment acupoints and completing study procedures remotely, 2) be assigned a treatment kit, 3) answer questions about their personal and health-related information for assessing their health condition before, during, and after the treatment during follow-up sessions, and 4) collect inner eyelid images for examining the hemoglobin level on a weekly basis at steady phase and daily basis during acute vaso-occlusive crisis stage.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* 14-17 (Adolescents) and 18-80 (Adults) years old
* Have been diagnosed with SCD and experiencing chronic pain in the past 6 months or vaso-occlusive crisis/crises in the past 12 months.
* Either outpatient or inpatient or status changing between each other
* Willing to limit the current and the introduction of any new medications or treatment modalities for control of pain symptoms during the study visits.
* Willing to stick to the scheduled acupressure treatments every other day for 5 weeks.
* Fluent in English and capable of giving written informed consent.

Exclusion Criteria:

* Recent/ongoing alternative pain management with acupuncture/acupressure or acupuncture/acupressure-related techniques within the last 6 months.
* Presence of a concurrent autoimmune or inflammatory disease such as rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, etc. that causes pain or any other chronic pain condition with pain greater than sickle pain.
* Diseases/conditions history includes but not limited to:
* Head injury with substantial loss of consciousness
* Known non-SCD-related severe psychiatric illnesses (e.g. current schizophrenia, major depression with suicidal ideation).
* Significant visual, motor, or auditory impairment that would interfere with ability to perform study visits-related activities

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Severity | Baseline and post-week 5 treatment
  Severity of pain will be assessed by Brief Pain Inventory (BPI) using the rating from 0= no pain to 10= worst pain imaginable.
Change in Pain Interference | Baseline and post-week 5 treatment
  Pain interference will be assessed by Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Questionnaire using the rating from with 4 = minimal interference to 20 = significant interference.

SECONDARY OUTCOMES:
Change in Nociplastic Pain Questionnaire | Baseline and post-week 5 treatment
  A customized questionnaire that is used to examine the locations (Yes/No) and severity of the pain interference (no problem-slight-moderate-severe) for understanding the level of nociplastic pain in the past 7 days. Widespread Pain Index and Symptom Severity will be scored from 0 to 10. Higher score connotes higher severity of nociplastic pain.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Questionnaire | Baseline and post-week 5 treatment
  Physical dysfunction, anxiety, depression, fatigue, sleep disturbance will be assessed by PROMIS-29, a single 4-20 numeric rating for each question.
Change in Multidimensional Fatigue Inventory (MFI) Questionnaire | Baseline and post-week 5 treatment
  MFI is a 20-item self-report instrument designed to measure fatigue with five dimensions including General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity. Subscale scores (range 4-20) are calculated as the sum of item ratings and a total fatigue score (range 20-100) is calculated as the sum of subscale scores. Higher scores indicate a higher level of fatigue.
Change in Pittsburgh Sleep Quality Index (PSQI) Questionnaire | Baseline and post-week 5 treatment
  The PSQI is a 19-item, self-rated questionnaire designed to measure sleep quality and disturbance over the past month in clinical populations. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
Change in Pediatric Quality of Life Inventory (PedsQL, both pediatric and adult versions) Questionnaire | Baseline and post-week 5 treatment
  The PedsQL is a self-report and parent-report measure assessing the quality of life in a variety of domains including physical, emotional, social, and school. Items are reverse-scored and transformed to a 0-100 scale where higher scores indicate better quality of life.
Change in opioid requirements | Baseline to 3 months post-treatment
  Opioid requirements will be assessed by morphine milligram equivalents.
Changes in vaso-occlusive crises (VOCs) frequency | Baseline and 6 months post-treatment
  The total number of VOCs within 6 months before and after the 5-week treatment will be documented.

OTHER OUTCOMES:
Blood Hemoglobin Level | Baseline, weekly through Week 5, and daily during VOCs up to 6 months
  Blood hemoglobin level will be assessed using self-collected images of the participants' inner eyelid via a patented algorithm of spectral super-resolution spectroscopy technique.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, Irvine, Irvine, California
  - Indiana University School of Medicine, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Houran L, Pucka AQ, Jiang M, Liu Z, O'Brien AR, Harte SE, Harris RE, Pakbaz Z, Wang Y. Acupressure alleviates pain and clinical symptoms in patients with sickle cell disease. medRxiv [Preprint]. 2025 May 1:2025.04.29.25326671. doi: 10.1101/2025.04.29.25326671. PMID 40343035